CLINICAL TRIAL: NCT03936296
Title: Comparison of Prostate Cancer Detection Rates of Standard Transrectal Prostate Biopsy and Multiparametric Prostate MR Guided MR-US Fusion Transrectal Prostate Biopsy
Brief Title: Prostate Cancer Detection Rates of Standard Transrectal Prostate Biopsy and MR-guided Fusion Transrectal Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Md, Assoc Prof, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TSG-2016-5200
Record Dates: First submitted 2019-04-30; First posted 2019-05-03 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: multiparametric prostate magnetic resonance imaging; MR-US fusion; MR guided prostate biopsy; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: To perform standard transrectal prostate biopsy and MR guided MR-US fusion prostate biopsy in the 2 randomized patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fusion arm (Active Comparator): Patients in this arm will be undertaken standard transrectal prostate biopsy and MR guided MR-US fusion prostate biopsy
  Interventions: Procedure: mpMR guided MR-US fusion transrectal prostate biopsy
- Standard arm (Other): Patients in this arm will be undertaken only standard transrectal prostate biopsy
  Interventions: Procedure: 12 core standard transrectal prostate biopsy

INTERVENTIONS:
Procedure: mpMR guided MR-US fusion transrectal prostate biopsy — mpMR images will be loaded to US fusion platform and registration of the will be performed. Suspicious lesions on MR which have PIRADS score 3 and above are targeted. Additional 2-4 cores biopsies will be taken them
  Other Names: Fusion biopsy
  Arms: fusion arm
Procedure: 12 core standard transrectal prostate biopsy — Under the guidance of transrectal ultrasonography, 12 core biopsies taken from apex, apex lateral, mid, mid lateral, base and base lateral of right and left prostate lobe
  Other Names: STRUS-B
  Arms: Standard arm

SUMMARY:
Prostate cancer is the most frequent cancer in men. Today serum prostate specific antigen (PSA) level and digital rectal examination (DRE) are routinely used for screening of prostate cancer. In the case of higher PSA levels and/or abnormal DRE, 10-12 core standard transrectal prostate biopsy (STRUS-B) is preferred method.Most of the pathological T1 stage tumours are diagnosed by this method. But as the prostate volume increases, cancer detection rate of STRUS-B decreases.In the last decade multiparametric prostate magnetic resonance imaging (mpMR) has gained importance in the diagnosis of prostate cancer beside the staging. Now it is possible to biopsies from lesions which are suspicious for cancer in mpMR. Recent studies have shown that mpMR guided prostate biopsies either transrectally or perineally have better cancer detection rates comparing STRUS-B, especially in patients with history of negative previous biopsy. But its use in biopsy naive settings is not recommended.In this study it is aimed to compare cancer detection rate of MR guided MR-US fusion transrectal prostate biopsy with STRUS-B.

DETAILED DESCRIPTION:
A histopathological evaluation of STRUS-B materials based on suspicious DRE findings and high or increasing PSA levels is the gold standard in prostate cancer diagnosis. However, the fact that approximately one-third of malignant prostate lesions is isoechoic and cannot be detected using conventional grayscale transrectal ultrasonography (TRUS) decreases the sensitivity rates of STRUS-B. These restrictions on the use of TRUS have encouraged urologists to use new methods to diagnose prostate cancer. One of these methods is the biopsy of lesions defined using mpMR, which has been widely used for the past 10 years. An MR targeted biopsy can be performed cognitively under MR guidance or using ultrasound devices with fusion software that can combine MR images with sonographic images. mpMR targeted biopsies are recommended in the current clinical practice for re-biopsies of patients who had previous negative biopsy but clinically suspected of cancer, follow-up biopsies of active surveillance, and biopsies of patients who are suspected to have recurrence after local minimally invasive treatment, such as radiotherapy and high-intensity focused ultrasonography. Recent studies showed that the cancer detection rate of mpMRIguided prostate biopsy is between 33.7% and 79.5%, which is higher than that of standard 12-core transrectal biopsy. However, the number of studies evaluating the use of MR targeted prostate biopsy in biopsy naive patients is limited.

In this study it is aimed to compare cancer detection rates of STRUS-B and MR guided MR-US fusion transrectal prostate biopsy in the biopsy naive patient setting.

100 patients will be randomized to STRUS-B arm and another 100 to fusion arm. In the standard arm patients who have high PSA levels and/or suspicious DRE will be undertaken STRUS-B. In the study arm all patients will undergo a multiparametric prostate MR without endorectal coils. MRI will be performed by Siemens Magnetom(Trade mark) 1.5 T (Siemens Medical Solutions, Pennsylvania, USA) MRI system. The images wi,ll be reviewed by an experienced uro-radiologist who has no detailed clinical information about the patients. Suspected areas in T2, T1 contrast, and diffusion-weighted images of multiparametric MRI were reported according to Prostate Imaging Reporting and Data System Version-2 (PIRADS v2). In cases of multiple lesions with different PIRADS scores, the lesion with the highest PIRADS score will be accepted as dominant lesion. Biopsy procedures will be performed under local anesthesia or sedoanalgesia. However, sedoanalgesia will be preferred if the patient could not tolerate pain during the penetration of US probe due to low pain threshold or anal canal stricture due to previous rectal surgeries. The procedure will be performed in outpatient clinic conditions. Transrectal ultrasonography will be performed by using an ultrasonography system with rigid fusion software (LOGIQ E9; General Electric, Massachusetts, USA) when patients lie on the left decubitus position. Rectal lidocaine gel will be applied 5 min before rectal US probe is introduced. A sonographic examination of the prostate tissue will be performed to check the presence of prominent lesions. Total prostate volumes will be measured. Multiparametric prostate MRI images will be uploaded to the US system on the day of biopsy. After segmentation (matching) of MRI images with sonographic images, the lesions reported in mpMR will be marked. The periprostatic block will be then performed with 2% prilocaine hydrochloride (20 mg/mL) injected into the neurovascular bundle on both sides of the prostate, with 5 mL to the right and 5 mL to the left. Following the block, two to five core biopsies from the MRI-targeted lesions with PIRADS ≥3 will be obtained. All procedures in fusion biopsy will be performed by two urologists experienced and trained in transrectal prostate ultrasonography and biopsy. After the F-TRUS biopsy completed, a standard 12-core TRUS biopsy will performed on fusion group. STRUS_B arm only standard 12 core transrectal prostate biopsy will be performed. A histopathological evaluation of biopsy specimens will be performed by a uro-pathologist with >10 years of experience. The percentage of cancer within the core, primary, and secondary Gleason score and grade according to the 2014 International Society of Urological Pathology (ISUP) grade will be specified in the final pathology report. Patients reported with high-grade prostatic intraepithelial neoplasm in three or more cores or atypical small acinar proliferation will be redirected to rebiopsy, but they will be included to the benign group in the evaluation of the present study.

As the secondary outcomes, pain level during MR fusion biopsy and STRUS biopsy evaluated by visual analogue scale score, cancer detection rates of different core numbers taken form MR targeted lesion, role of the peripheric blood parameters (such as, neutrophil to lymphocyte ratio and systemic immune inflammatuary index) in predicting prostate cancer in PRIADS 3,4 and 5lesions, and comparison of the tumor laterality and ISUP grade in MR US fuison biopsy and radical prostatectomy specimens will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

PSA level 2,5-10mg/dl Approving the transrectal prostate biopsy and mpMR NO contraindication for MR: glomerular filtration rate (GFR) >60ml/dk, no claustrophobia, no prosthesis or cardiac pacemaker which is not suitable for MR no contraindication for stopping antiaggregant or antithrombotic treatment. no history of previous prostate biopsy no diagnosis of prostate cancer or other malignancies

Exclusion Criteria:

* not approving the biopsy and MR imaging
* having prosthesis or cardiac pace maker not suitable for MR
* having contraindication for stopping antiaggregant or antithrombotic treatment.
* history of previous prostate biopsy

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
cancer detection rate of MR-US fusion biopsies | 15 days after biopsy
  percentage of prostate cancer detected by fusion biopsies
clinically significant cancer detection rate of MR-US fusion biopsies | 15 days after biopsy
  percentage of prostate cancer which is ISUP group 2 and above detected by fusion biopsies
cancer detection rate of STRUS-B | 15 days after biopsy
  percentage of prostate cancer detected by STRUS-B
clinically significant cancer detection rate of STRUS-B | 15 days after biopsy
  percentage of prostate cancer which is ISUP group 2 and above detected by STRUS-B
cancer detection rate of combined method (fusion + STRUS-B ) | 15 days after biopsy
  percentage of prostate cancer detected by combined method
clinically significant cancer detection rate of combined method (fusion + STRUS-B ) | 15 days after biopsy
  percentage of prostate cancer which is ISUP group 2 and above detected by combined method

SECONDARY OUTCOMES:
Visual analogue Scale score for pain | Just after the biopsy
  To score the pain level that expreinced by patients during STRUS-B and MR-US bx
Comparison of the cancer detection rate of different core numbers taken from MR lesion. | 15 days after biopsy
  Cancer detection rate of the 2, 3 and 4 cores taken from PIRADS 3,4 and 5 lesion
Neutrophil to lymphocyte ratio to predict cancer in different PRIADS lesions. | 15 days after biopsy
  Neutrophil to lymphocyte ratio to predict cancer in different PRIADS lesions.
Role of Systemic immune-infllamatuary index to predict the caner in PIRADS 3,4 5 lesions | 15 days after biopsy
  neutrophil x platelet count /lymphocyte count
Tumor upgrade rate of MR US fusion biopsy in radical prostatectomy specimens | 15 days after radical prosatetctomy
  comparison of the ISUP grade of MR-fusion biopsy and radical prostatectomy speimens at whom underwent radical prostatectomy
Tumor laterality in biopsy specimens and radical prostatectomy specimens | 15 days after radical prosatetctomy
  Tumor laterality in biopsy specimens and radical prostatectomy specimens

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demritas, Assoc Prof, Principal Investigator — Erciyes University Faculty of Medicine
Locations (1):
- Department of Urology, Ercieys University, Faculty Of Medicine,, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durmus T, Baur A, Hamm B. Multiparametric magnetic resonance imaging in the detection of prostate cancer. Aktuelle Urol. 2014 Mar;45(2):119-26. doi: 10.1055/s-0034-1371875. Epub 2014 Apr 3. PMID 24700068
- [Background] Hong CW, Amalou H, Xu S, Turkbey B, Yan P, Kruecker J, Pinto PA, Choyke PL, Wood BJ. Prostate biopsy for the interventional radiologist. J Vasc Interv Radiol. 2014 May;25(5):675-84. doi: 10.1016/j.jvir.2013.12.568. Epub 2014 Feb 26. PMID 24581731
- [Background] Liao S, Gao Y, Oto A, Shen D. Representation learning: a unified deep learning framework for automatic prostate MR segmentation. Med Image Comput Comput Assist Interv. 2013;16(Pt 2):254-61. doi: 10.1007/978-3-642-40763-5_32. PMID 24579148
- [Background] Epstein JI, Egevad L, Amin MB, Delahunt B, Srigley JR, Humphrey PA; Grading Committee. The 2014 International Society of Urological Pathology (ISUP) Consensus Conference on Gleason Grading of Prostatic Carcinoma: Definition of Grading Patterns and Proposal for a New Grading System. Am J Surg Pathol. 2016 Feb;40(2):244-52. doi: 10.1097/PAS.0000000000000530. PMID 26492179
- [Background] Barentsz JO, Weinreb JC, Verma S, Thoeny HC, Tempany CM, Shtern F, Padhani AR, Margolis D, Macura KJ, Haider MA, Cornud F, Choyke PL. Synopsis of the PI-RADS v2 Guidelines for Multiparametric Prostate Magnetic Resonance Imaging and Recommendations for Use. Eur Urol. 2016 Jan;69(1):41-9. doi: 10.1016/j.eururo.2015.08.038. Epub 2015 Sep 8. No abstract available. PMID 26361169
- [Result] Kuru TH, Roethke MC, Seidenader J, Simpfendorfer T, Boxler S, Alammar K, Rieker P, Popeneciu VI, Roth W, Pahernik S, Schlemmer HP, Hohenfellner M, Hadaschik BA. Critical evaluation of magnetic resonance imaging targeted, transrectal ultrasound guided transperineal fusion biopsy for detection of prostate cancer. J Urol. 2013 Oct;190(4):1380-6. doi: 10.1016/j.juro.2013.04.043. Epub 2013 Apr 19. PMID 23608676
- [Result] Pokorny MR, de Rooij M, Duncan E, Schroder FH, Parkinson R, Barentsz JO, Thompson LC. Prospective study of diagnostic accuracy comparing prostate cancer detection by transrectal ultrasound-guided biopsy versus magnetic resonance (MR) imaging with subsequent MR-guided biopsy in men without previous prostate biopsies. Eur Urol. 2014 Jul;66(1):22-9. doi: 10.1016/j.eururo.2014.03.002. Epub 2014 Mar 14. PMID 24666839
- [Result] Junker D, Schafer G, Heidegger I, Bektic J, Ladurner M, Jaschke W, Aigner F. Multiparametric magnetic resonance imaging/transrectal ultrasound fusion targeted biopsy of the prostate: preliminary results of a prospective single-centre study. Urol Int. 2015;94(3):313-8. doi: 10.1159/000365489. Epub 2015 Jan 9. PMID 25591786
- [Result] Abd-Alazeez M, Kirkham A, Ahmed HU, Arya M, Anastasiadis E, Charman SC, Freeman A, Emberton M. Performance of multiparametric MRI in men at risk of prostate cancer before the first biopsy: a paired validating cohort study using template prostate mapping biopsies as the reference standard. Prostate Cancer Prostatic Dis. 2014 Mar;17(1):40-6. doi: 10.1038/pcan.2013.43. Epub 2013 Oct 15. PMID 24126797
- [Result] Delongchamps NB, Peyromaure M, Schull A, Beuvon F, Bouazza N, Flam T, Zerbib M, Muradyan N, Legman P, Cornud F. Prebiopsy magnetic resonance imaging and prostate cancer detection: comparison of random and targeted biopsies. J Urol. 2013 Feb;189(2):493-9. doi: 10.1016/j.juro.2012.08.195. Epub 2012 Oct 8. PMID 22982424
- [Derived] Sonmez G, Demirtas T, Tombul ST, Ozturk F, Demirtas A. What is the ideal number of biopsy cores per lesion in targeted prostate biopsy? Prostate Int. 2020 Sep;8(3):112-115. doi: 10.1016/j.prnil.2020.03.004. Epub 2020 Apr 23. PMID 33102391